CLINICAL TRIAL: NCT02276638
Title: Comparative Study of the Specular Microscopes for Center Point Method and Corner Point Method for the Measurements of Endothelial Cell Density Measurements, Coefficient of Variation of Endothelial Cell Area and % Hexagonality.
Brief Title: Comparative Study of Specular Microscopes for Measurements of Cell Density, Coefficient of Variation and Hexagonality
Status: Completed | Type: Observational
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: CEM-530-US-0002
Record Dates: First submitted 2014-10-14; First posted 2014-10-28 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Corneal Endothelial Cell Loss
MeSH Terms: conditions — Corneal Endothelial Cell Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 18-28 years old Non-pathologic: Device: Specular Microscope Nidek CEM-530 Device: Specular Microscope Konan CELLCHEK XL
  Interventions: Device: Specular Microscope Nidek CEM-530; Device: Specular Microscope Konan CELLCHEK XL
- 29-80 years old Non-pathologic: Device: Specular Microscope Nidek CEM-530 Device: Specular Microscope Konan CELLCHEK XL
  Interventions: Device: Specular Microscope Nidek CEM-530; Device: Specular Microscope Konan CELLCHEK XL
- 29-80 years old pathological: Device: Specular Microscope Nidek CEM-530 Device: Specular Microscope Konan CELLCHEK XL
  Interventions: Device: Specular Microscope Nidek CEM-530; Device: Specular Microscope Konan CELLCHEK XL

INTERVENTIONS:
Device: Specular Microscope Nidek CEM-530 — Nidek CEM-530
Device: Specular Microscope Konan CELLCHEK XL — Konan CELLCHEK XL

SUMMARY:
The primary objective of this clinical study is to collect clinical data to support an FDA 510(k) submission for the Nidek CEM-530 Center point method and Corner point method. The secondary objective is to evaluate any adverse events found during the clinical study.

DETAILED DESCRIPTION:
The primary objective of this clinical study is to collect clinical data to support an FDA 510(k) submission for the Nidek CEM-530 Center point method and Corner point method.

ELIGIBILITY:
Inclusion Criteria:

* Non-Pathologic: Male or female subjects from 18 to 80 years old who have full legal capacity to volunteer on the date the informed consent is signed. Subjects who can follow the instructions by the clinical staff at the clinical site,and can attend examinations on the scheduled examination date. Subjects who agree to participate in the study.
* Pathologic: Male and female subjects from 29 to 80 years old who have full legal capacity to volunteer on the date the informed consent is signed. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date. Subjects who agree to participate in the study. At least one eye with any of the following conditions:

  * History of post-op surgical trauma including bullous keratopathy
  * History of corneal transplant
  * Physical injury or trauma to the cornea
  * Long term Fuch's dystrophy, Guttata or other corneal endothelial dystrophies
  * Keratoconus
  * Long term PMMA contact lens use (greater than 3 years)

Exclusion Criteria:

* Non-Pathologic: Male and female subjects from 29 to 80 years old who have full legal capacity to volunteer on the date the informed consent is signed. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date. Subjects who agree to participate in the study. At least one eye with any of the following conditions:

  * History of post-op surgical trauma including bullous keratopathy
  * History of corneal transplant
  * Physical injury or trauma to the cornea
  * Long term Fuch's dystrophy, Guttata or other corneal endothelial dystrophies
  * Keratoconus
  * Long term PMMA contact lens use (greater than 3 years)
* Pathologic: History of cataract, refractive or ocular surgical procedures that render the cornea opaque or otherwise impact its ability to be imaged using the investigational device. Fixation problems which may prevent obtaining at least poor quality (refer to Figure 1) CEM-530 and KONAN CELLCHEK PLUS images in either eye.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ophthalmology Practice
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Andover Eye Associates
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 18-28 Years Old Non-pathologic: 18-28 years old Non-pathologic Device: Nidek CEM-530
- 29-80 Years Old Non-pathologic: 29-80 years old Non-pathologic Device: Nidek CEM-530
- 29-80 Years Old Pathological: 29-80 years old pathological Device: Nidek CEM-530
Period: Overall Study
Arm/Group | 18-28 Years Old Non-pathologic | 29-80 Years Old Non-pathologic | 29-80 Years Old Pathological
Started | 28 | 28 | 23
Completed | 28 | 28 | 23
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 18-28 Years Old Non-pathologic | 29-80 Years Old Non-pathologic | 29-80 Years Old Pathological | Total
Number analyzed (Participants) | 28 | 28 | 23 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 28 | 23 | 79
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.2 (3.8) | 53 (13.42) | 63.9 (12.39) | 44.1 (20.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 15 | 47
  Male | 15 | 9 | 8 | 32
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 23 | 79

OUTCOME MEASURES:

1. Primary Outcome: Center Method Corneal Endothelial Cell Density
Time Frame: single time point - 1 day
Population: Not all participants indicated in the Participant Flow Module were analysed.
Measure: Mean (Standard Deviation); unit: cells/mm2
Arm/Group | 18-28 Years Old Non-pathologic | 29-80 Years Old Non-pathologic | 29-80 Years Old Pathological
Number analyzed (Participants) | 28 | 27 | 19
cells/mm2 | 3069.5 (346.41) | 2678.6 (391.33) | 2514 (351.02)

2. Primary Outcome: Center Method Coefficient of Variation of Endothelial Cell Area
Description: Coefficient of variation(CV) is that Standard deviation (SD) divided by the average area of endothelial cell analyzed
Time Frame: single time point - 1 day
Population: Not all participants indicated in the Participant Flow Module were analysed.
Measure: Mean (Standard Deviation); unit: percent of Coefficient of variation
Arm/Group | 18-28 Years Old Non-pathologic | 29-80 Years Old Non-pathologic | 29-80 Years Old Pathological
Number analyzed (Participants) | 28 | 27 | 19
percent of Coefficient of variation | 20.3 (1.90) | 23.3 (3.27) | 23.0 (4.11)

3. Primary Outcome: Percentage Hexagonality
Description: Percentage hexagonality(%HEX) is that Proportion of hexagonal cells found in the analyzed endothelium
Time Frame: single time point - 1 day
Population: Not all participants indicated in the Participant Flow Module were analysed.
Measure: Mean (Standard Deviation); unit: Percentage hexagonality
Arm/Group | 18-28 Years Old Non-pathologic | 29-80 Years Old Non-pathologic | 29-80 Years Old Pathological
Number analyzed (Participants) | 28 | 27 | 19
Percentage hexagonality | 63.0 (6.33) | 57.1 (6.66) | 58.7 (7.96)

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- 18-28 Years Old Non-pathologic; 29-9- Years Old Non-pathologic; 29-80 Years Old Pathological: Device: Nidek CEM-530 Device: Konan Specular Microscope CELLCHEK XL
  Specular Microscope: Nidek CEM-530
  Specular Microscope: Konan CELLCHECK XL
Arm/Group | 18-28 Years Old Non-pathologic | 29-9- Years Old Non-pathologic | 29-80 Years Old Pathological
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/23
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No